CLINICAL TRIAL: NCT06593262
Title: Efficacy of Digital Cognitive Behavioral Therapy for Insomnia (CBT-I) with Artificial Intelligence Chatbot for Youth with Insomnia: an Assessor-blind, Randomized Controlled Trial
Brief Title: Efficacy of Digital Cognitive Behavioral Therapy for Insomnia (CBT-I)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tim M. H. Li, Prof., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14106223
Record Dates: First submitted 2024-08-18; First posted 2024-09-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- app-based digital cognitive behavioral therapy for insomnia with AI chatbot (Experimental)
  Interventions: Behavioral: app-based digital cognitive behavioral therapy for insomnia with AI chatbot
- app-based digital cognitive behavioral therapy for insomnia without AI chatbot (Active Comparator)
  Interventions: Behavioral: app-based digital cognitive behavioral therapy for insomnia without AI chatbot

INTERVENTIONS:
Behavioral: app-based digital cognitive behavioral therapy for insomnia with AI chatbot — digital cognitive behavioral therapy for insomnia with two-way interactive, intelligent, and patient-centered conversational agents
  Arms: app-based digital cognitive behavioral therapy for insomnia with AI chatbot
Behavioral: app-based digital cognitive behavioral therapy for insomnia without AI chatbot — digital cognitive behavioral therapy for insomnia without two-way interactive, intelligent, and patient-centered conversational agents
  Arms: app-based digital cognitive behavioral therapy for insomnia without AI chatbot

SUMMARY:
Insomnia is a common sleep problem, which affects 9.4-38.2% of youths worldwide. Youth insomnia is linked to mental health problems, leading to substantial health and economic burden. The project aims to conduct an assessor-blind, randomized controlled trial to evaluate the efficacy of an app-based CBT-I with AI chatbot in reducing insomnia symptoms among youths, compared to an app-based CBT-I without AI chatbot.

ELIGIBILITY:
Inclusion Criteria:

i. Youth aged 18 to 25 years (as defined by WHO and evidence on AI mental health chatbots only available for individuals aged 18 years and older)

ii. Online informed consent of participation in the study should be provided

iii. Willing to comply with the requirements of the study protocol

iv. The presence of moderate to severe insomnia measured by a score of 15 or above on the Insomnia Severity Index (ISI)

v. difficulties initiating, maintaining or nonrestorative sleep over a 1-month period

vi. Having access to a smartphone and consistent internet access for their smartphone

vii. Accepting the terms of service and privacy policies of the mobile apps used in the study for the delivery of the intervention

Exclusion Criteria:

i. A history of any sleep disorder(s) (other than insomnia disorder) such as narcolepsy, obstructive sleep apnea, and restless legs syndrome

ii. A history of any mental retardation or neuropsychiatric disorder(s) (other than depression and anxiety disorders as they are the secondary outcomes) such as bipolar disorder, schizophrenia, and substance use disorder

iii. Presence of serious suicidality as evidenced by ideation with a plan or an attempt

iv. Receiving any pharmacological treatment (including sleep promoting agents)

v. Receiving any structured psychotherapy

vi. Having shiftwork and trans-meridian travel in the past 3 months and during the intervention

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | a) baseline; b) interim during intervention (2-week after baseline); c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  the severity of insomnia symptoms

SECONDARY OUTCOMES:
sleep onset latency (SOL) | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  7-day sleep diary
wake after sleep onset (WASO) | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  7-day sleep diary
sleep efficiency (SE) | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  7-day sleep diary
Total sleep time (TST) | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  7-day sleep diary
The Pre-Sleep Arousal Scale | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  cognitive and somatic manifestations of arousal near bedtime Total score ranges from 8 to 40. Higher scores suggest increased cognitive and somatic arousal before sleep.
The Cognitive Failures Questionnaire | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  self-reported failures in perception, memory, and motor function Total score ranges from 0 to 100. Higher scores indicate more self-reported cognitive lapses.
Ford Insomnia Response to Stress Test | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  personal vulnerability to stress-related insomnia Total score ranges from 9 to 36. Higher scores suggest a greater likelihood of stress-induced insomnia.
reduced Horne and Östberg Morningness and Eveningness Questionnaire | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  Chronotype preference. Total score ranges from 4 to 25. Higher scores suggest a morning chronotype, while lower scores indicate an evening chronotype.
The Dysfunctional Beliefs and Attitudes about Sleep Scale | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  Faulty sleep-related beliefs and cognitions, which are cognitive aspects typically involved in the maintenance of insomnia. Total score range of 0 to 160, with higher scores indicating stronger dysfunctional beliefs about sleep.
Patient Health Questionnaire-9 | a) baseline; b) interim during intervention (2-week after baseline); c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  The severity of depressive symptoms. Total score range of 0 to 27, where higher scores signify higher levels of depressive symptoms.
General Anxiety Disorder-7 | a) baseline; b) interim during intervention (2-week after baseline); c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  The severity of anxiety symptoms. Total score range of 0 to 21, with higher scores reflecting higher levels of anxiety symptoms
The Sleep Hygiene Index | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  The practice of sleep hygiene behaviors. Total score ranges from 0 to 52. Higher scores reflect poorer sleep hygiene practices.
The Charlotte Attitudes Towards Sleep Scale | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  Perception and attitude towards sleep in youths. Total averaged score ranges from 1 to 7. Higher scores denote more positive attitudes about sleep.
The Multidimensional Fatigue Inventory | a) baseline; c) post-intervention (1-month after baseline); d) 3-month after intervention (4-month after baseline); e) 6-month after intervention (7-month after baseline)
  Five dimensions of fatigue (general fatigue, physical fatigues, mental fatigue, decreased motivation, and decreased activities).
  Total score ranges from 20 to 100. Higher scores indicate greater fatigue levels.

OTHER OUTCOMES:
Treatment Satisfaction Scale | post-intervention (1-month after baseline)
  Treatment Satisfaction Scale includes 8 items with 5-point Likert scale. The total score ranges from 8 to 40. The higher the score means a higher satisfaction.
Treatment Component Adherence | post-intervention (1-month after baseline)
  Treatment Component Adherence Scale. 26 single-item, each item has a scoring between 1 to 5.
Acceptability E-scale questionnaire | post-intervention (1-month after baseline)
  Measures the digital program was acceptable or not. Total scores range from 6 to 30. The higher the score means a more positive evaluation.
The Embodied Conversational Agents Trust Questionnaire | post-intervention (1-month after baseline)
  Measures trust towards the mHealth technologies. Total score ranges from 0 to 15. Higher scores indicate a more positive attitude or greater trust towards the mHealth agent or technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided